CLINICAL TRIAL: NCT02722226
Title: The Impact of a High Fidelity Simulation Based Sedation Training on the Performance of Non-anesthesiologists Residents for the Management of Complications Associated to Sedation.
Brief Title: High Fidelity Simulation and Sedation Training of Non-anesthesiologists Residents
Acronym: DedSim
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Issam Tanoubi (Other)
Responsible Party: Sponsor-Investigator, Issam Tanoubi, MD, Assistant Professor, Université de Montréal
Organization: Université de Montréal (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SedSim1
Record Dates: First submitted 2016-03-17; First posted 2016-03-29 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Performance of Non-anesthesiologists Residents for the Management of Sedation's Complications
Keywords: High fidelity simulation; Sedation; Medical education
MeSH Terms: interventions — Airway Management; Crew Resource Management, Healthcare

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simulation based sedation learning (Intervention Group) (Experimental): The program includes online learning. It is followed by development of interactive presentations, based on simulated cases or simulated patients (actors), low fidelity simulation for specific technical skills as well as high fidelity scenarios of complications related to sedation.
  Interventions: Other: Simulation; Device: Airway management; Behavioral: Crisis resource management
- Control Group (No Intervention)

INTERVENTIONS:
Other: Simulation — High fidelity simulation based sedation learning program
  Arms: Simulation based sedation learning (Intervention Group)
Device: Airway management — Workshop on using airway management and oxygenation devices.
  Arms: Simulation based sedation learning (Intervention Group)
Behavioral: Crisis resource management — Learning crisis resource management principles
  Arms: Simulation based sedation learning (Intervention Group)

SUMMARY:
Objective Sedation is a depression of consciousness varies between anxiolysis and general anesthesia. It is used to facilitate diagnostic tests and minor surgeries. Respiratory complication is the main side effect of the sedation. His Early diagnosis and adequate management prevent serious complications such as hypoxic brain damage or death. A development of a learning program of sedation is required. Simulation as a teaching tool has improved the clinical expertise of learners. The objective of the study is to evaluate the impact of a simulation based medical education program on the performance of non-resident anesthesiologists for the management of complications related to sedation.

Methods This trial is randomized, controlled and single blinded. Non-resident anesthesiologists, without prior training on sedation, are included and randomized to receive or not a simulation based sedation learning. This program includes a pharmacology sedatives learning, teaching technical skills for airway management on low fidelity mannequin and high-fidelity simulation scenarios of these complications. Two evaluators, single-blinded, visualise the recorded performance of residents in simulation session. The evaluation is based on a performance checklist developed by Delphi technique. It compares the performance of the residents within the same group before and after the simulation based medical education program and to compare groups of residents.

Data analysis The sample size is based on similar simulation studies. The results are compared with the variance analysis for repeated measures. The difference in performance before and after simulation is compared using a t test.

The investigators hypotheses that improved performance scores following the simulation based medical education would put the dot on the importance of simulation as a learning tool.

DETAILED DESCRIPTION:
Sedation is a drug depression of consciousness and alertness. It involves intravenous hypnotics and narcotics administration. Depending on doses and blood levels of administered agents, there is a continuum between anxiolysis, light sedation (monitored anesthesia care), deep sedation and general anesthesia.

Sedation is used to facilitate diagnostic examinations, minor surgery, endoscopic surgery and endovascular or transcutaneous therapeutic radiological procedures. It provides comfort to the patient during the procedure and better conditions for examination or treatment for the operator.

The main risk during procedural sedation is compromising the patient's respiratory function and airway. The obstruction of the upper airway by the tongue, soft palate or epiglottis on one hand and respiratory depression due to the sedative on the other hand are the major problems of sedation. In addition to respiratory depression, decreased airway protective reflexes during sedation exposes to the gastric contents aspiration and consequent respiratory complications.

Major complications are rare: one case of death of 160,000, 1 case of tracheal intubation of 58 000 and no cases of permanent neurologic damage of 646,000 gastrointestinal endoscopies performed under sedation. More common, the incidence of partial obstructions requiring airway maneuvers release (mandibular subluxation, oropharyngeal airway device, nasopharyngeal airway device) is 14.4%, 12.8% of hypoxemia, 0.1% of ventilation with face mask and in 0.6% the ongoing procedure needed to be stopped.

Although these incidents are without clinical severity, they can cause serious complications if diagnosed late or in inadequate care. Various analyzes of the American Society of Anesthesiology claims related to sedation, prove the seriousness of these complications and the importance of their early management, 40% of claims involving death or hypoxic permanent brain injury could be prevented and 50% of claims are related to anesthetic procedures performed outside the operating room. Respiratory depression associated with an absolute or relative overdose of sedative is the primary mechanism of complications.

Sedation can be practiced by non-anesthesiologists. There are several publications, other than in the anesthesiology field, on sedation regimes used and their safety and efficacy. The heterogeneity of definitions of respiratory complications and lack of power of these studies failed to show a reduction in respiratory complications and safety of sedation according to the standards of the anesthesiologist. The complications are associated to limited knowledge of anesthetic drugs pharmacology, the monitoring of sedation and the airway management. The anesthesiologist should play a central role in establishing safe sedation standards when administered by non-anesthesiologists.

In addition to the sedation learning need, the majority of residents and non-anesthesiologists sedation practitioners, strongly express their interest in a learning sedation. This interest is related to the residents' discomfort when using sedation associated to a lack of mastering of sedatives pharmacology and airway managements principles.

The simulation as a teaching tool is increasingly used. The literature has shown that simulation can improve the performance of trainees in various technical and non technical skills (expertise, crisis resource management principles).

Simulation is used as an assessment tool of education techniques. It assesses the performance of trainees through reproducible situation.

Simulation based medical education success depends on several factors. The relevance of the subject taught in the professional context, the target population, the identification of educational goals, the educational activities implemented to achieve these objectives, the choice of parameters to be measured and the measurement method are all factors that can strongly affect the impact of the simulation based medical education.

The recent meta-analysis of McGraphie and colleagues reviewed all the studies, from 1990 to 2011, evaluating the effectiveness of simulation based medical education. It shows the simulation based medical education superiority over the traditional clinical education in acquiring limited designed skills. The explanation of simulation use is based on the fact that the simulation seems to fill some gaps of traditional clinical learning, such as delayed and random clinical exposure and scarcity of complications.

The use of simulation for learning sedation to non-anesthesiologists seems to meet the requirements dictated by the subject to teach. It should, indeed, allow sedative drugs pharmacology learning and technical skills mastering. It should also allow, through reproducible scenarios, in high-fidelity simulation, improvement of the overall complications' sedation management and the assessment of the impact of simulation based medical education. However, even if the simulation offers all the theoretical and practical components of safe sedation educational program, the overall result of education based on simulation on the ability of non-resident anesthesiologists to manage sedation's complications remains to be assessed.

The aim of this randomized controlled trial is to evaluate the impact of a high fidelity simulation based sedation learning on non-anesthesiologists residents' performance in the management of sedation's complications, during simulated scenarios.

Methods

1. Description of the simulation based sedation learning program

   The program's goal is to offer a comprehensive approach to theory and practice of sedation. It must provide the resident a vision adapted to their daily practice. Being based on the simulation, education should draw profile of all components provided to education from simulation tool.

   The simulation based sedation learning program consists of different modules in response to residents' needs in the practice of sedation. The teaching is based on specific educational objectives, experimental learning conditions, repeated practice and an assessment based on the achievement rate of tasks. These modules are developed by anesthesiologists practicing in academic fields and practicing sedation.

   The program includes online learning. It is followed by development of interactive presentations, based on simulated cases or simulated patients (actors), low fidelity simulation for specific technical skills as well as high fidelity scenarios of complications related to sedation. The purpose of the high-fidelity simulation is to enable the resident to integrate theoretical and practical learning received, in a similar context to his clinical practice, to develop a comprehensive and contextual (material, human resources and authorized techniques) management of sedation, to prevent, to anticipate, to make an early diagnosis and adequate management of simulated complications.
2. Study Design

   This is a prospective, randomized, controlled, single-blind, trial. The study is conducted in the University of Montreal simulation centre. The robotic model used is the SimMan 3G (Laerdal, Inc. http: / /www.laerdal.com/doc/85/SimMan-3G).

   The primary objective is the performance scores before and after a simulation based sedation learning program during a high fidelity simulated scenario of sedation's complications managed by non anesthesiologists residents.
3. Population Included in this study, all residents from surgery programs, radiology, gastroenterology, pneumology, family medicine , emergency medicine of the University of Montreal. Residents must have academic supervision with 1: 1 by a senior during their practice. Residents who have received prior instruction on sedation or advanced learning technical skills for airway management during residency will be excluded.

   The recruited participants were randomized according to a randomization table, computerized, established prior to inclusion in intervention group that receives simulation based sedation learning and control group.
4. Assessment method and developing the performance checklist The evaluation is based on a list of tasks and behaviours (technical and non technical skills) of the resident during the management of simulated complications related to sedation. It includes items related to the specific management of complications (expertise) and non-specific items of communication and collaboration (Crisis Resource Management principles). It is divided in a) an initial assessment of the situation b) diagnostic steps c) management d) secondary evaluation. The performance list is developed and validated using the modified Delphi method.
5. Procedure A description of the high-fidelity simulation is performed, and a participation in an uncomplicated sedation scenario is made initially for the two groups. This first experience allows them to become familiar with the environment of the simulation and the use of mannequin interface / physician. This simulation is not followed by a debriefing.

Participants are then randomized in:

Intervention group:

Residents included in this group will go through the following steps:

A simulation of respiratory complications related to sedation: Base line performance.

The simulation based sedation program, described above. A second simulation of respiratory complications related to sedation: Post test.

Assessments are conducted by independent instructors blindly. The evaluators attribute scores by viewing the recorded performances, without knowing the group to which the candidate is included, or whether simulation based sedation program is realized or not.

Control group:

Residents included in this group carry out:

A complication related to sedation simulation: Base line performance, not followed by a debriefing.

A self visualization of a video describing sedation in adults. A second simulation, about 2 months later: Post test For equity training, the control group will be offered the simulation based sedation program after the end of the study, if desired.

6. Analysis of results The tasks are classified in 2 categories: properly performed or not / not properly performed.

The performance score represents adequately performed tasks on the total number of tasks (primary outcome).

Secondary outcomes include the comparison of (a) performance scores between pre-test and post-test for each group (b) performance scores related to technical skills (c) performance scores related to non technical skills.

The results are compared with the analysis of variance for repeated measures. The difference in performance before and after the simulation based sedation program is compared using a t test.

The number of participants was the number of eligible residents and who agreed to participate (convenience sample). As the selected population in this study consists of a larger sample, as several residency programs are concerned, the investigators opt for two groups of 25 participants (total n 50).

ELIGIBILITY:
Inclusion Criteria:

* Residents from surgery programs, radiology, gastroenterology, pneumology, family medicine, emergency medicine of the University of Montreal
* Residents with academic supervision with 1: 1 by a senior during their clinical practice

Exclusion Criteria:

* Resident with prior instruction on sedation or advanced learning technical skills for airway management.
* Refusal to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-03; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Improved residents performance after simulation based education, measured by previously built performance grid | 3 to 6 months

REFERENCES:
- [Derived] Evain JN, Do T, Harkouk H, Drolet P, Perron R, Georgescu M, Robitaille A, Tanoubi I. Mastering Sedation and Associated Respiratory Events through Simulation-Based Training: A Randomised Controlled Trial Involving Non-Anaesthesiology Residents. Eur J Investig Health Psychol Educ. 2024 Feb 23;14(3):463-473. doi: 10.3390/ejihpe14030031. PMID 38534892